CLINICAL TRIAL: NCT04290169
Title: Utilizing Motion Controlled Video Games and Botulinum Toxin A Treatment to Improve Motor Function, Activity and Participation in Persons With Spastic Cerebral Palsy - a Single-subject Design Study
Brief Title: Effect of Video Game-assisted and BoNT-A Injection Therapy on Spasticity, Activity and Participation in CP Patients
Acronym: CPSpast
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Göteborg University (Other); CP-foreningen (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPSpast
Record Dates: First submitted 2020-02-17; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral palsy; Cognition; Spasticity; BoNT-A; Botulinum Toxin A; video game; balance; Upper extremity function
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: The single subject design was chosen due to its sensitivity to individual differences which is a relevant feature when studying heterogenous population as adults with spastic CP. The study is a multiple-treatment design with two intervention phases, an ABACAA design. The study include a baseline assessment phase (A1), a three-month intervention phase with motion controlled video game training (B), post-intervention assessment (A2), a second three-month intervention phase with Motion Controlled Video Game (MCVG) treatment and BoNT-A treatment (C) including an assessment in the middle when BoNT-A usually have its peak (6 weeks after application) (A3), post-intervention assessment three months after application of BoNT-A (A4) and a follow-up assessment 9 months after beginning of first intervention (A5). All participants will be medically examined and assessed with functional measures in all assessment phases. The timeframe from baseline to follow-up is approximately 9 months.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adults with hemiplegic spastic cerebral palsy (Other): Adults (> 18 years old) with hemiplegic spastic cerebral palsy, with reduced hand function and spasticity as prevalent finding under clinical examination. Also these patients can walk but have problems with balance. Participants' cognitive function does not limit them to perform video game training.
  Interventions: Drug: IncobotulinumtoxinA; Device: Video game

INTERVENTIONS:
Drug: IncobotulinumtoxinA — IncobotulinumtoxinA will be injected in upper extremities according to recommended guidelines. Two methods will be used in the study: auditive electromyography (EMG) and ultrasound guided injection technique. The decision process of which muscles to inject will be based on information obtained through examination of hand function, the presence of increased muscle tone during the clinical examination as well as a positive response from auditive EMG
  Other Names: Botulinum Toxin A, Xeomin, BoNT-A
Device: Video game — The study will include the Nintendo Switch or similar consoles that include games that require the players to move their bodies while holding motion controllers in order to progress. The games included in this project has been chosen by staff at our hospitals Virtual Gaming Lab. The participants are recommended to train 30 minutes each day, 4 days a week, during the training periods. It is expected that the amount of training will vary among the participants. Thus, each participant will be instructed to keep a training-diary and weekly report number of hours played/trained through an online reporting system created with "online form", an electronic data collection system available through the University of Oslo

SUMMARY:
Cerebral palsy (CP) is a non-progressive condition of the central nervous system caused by immature brain damage before, during or after birth. Persons affected by CP experience disability of various types. In individuals with CP, one of the most frequent symptoms is limited hand function. Other issues that often occur are muscle weakness, spasticity and problems with balance.

Injection with Botulinum Toxin A (BoNT-A) is common treatment for spasticity in patients with injury in central nervous system, e.g. traumatic brain injury, stroke, spinal cord injuries and CP.The main goal of the project is to explore if motion controlled video game treatment alone or in combination with injection treatment with BoNT-A lead to improvement of hand function, activity and participation in adults with CP.

In the project, the investigators will evaluate if these two interventions improve balance in adults with CP.

Participants will be psychologically tested in the beginning and the end of the project to evaluate if interventions can have positive effect on psychological symptoms such as depression and anxiety, The project is multidisciplinary. It involves a doctor, a nurse, an occupational therapist, a physiotherapist and a psychologist. The team will in ordinary clinical practice examine participants. Individual goals will be set up in agreement with each participant. The goals will be measurable, achievable and time bound. By reviewing scope of agreed goals, the investigators will be able to summarize most frequent problems that CP patients experience in their daily life.

There will be 25 participants in the study and they will be followed for 9 months. During every visit the team will examine participants, perform relevant tests and obtain objective and subjective outcomes. It will be assessed to what degree the goals have been achieved.

The investigators also want to evaluate long term effects of the two intervention applied in the study. Therefore, the participants will be finally assessed 3 months after last intervention period.

Based on study results, implications for future treatment volume and organization of the rehabilitation for persons with spasticity will be discussed with the participating units, hospitals, municipalities and policy makers. Professionals included in this project are also clinicians and will have an important role in ensuring that the findings are included in clinical guidelines and educational activities.

ELIGIBILITY:
Inclusion Criteria:

* Adults with CP (>= 18 years)
* Spastic CP with one upper extremity affected
* Grasp function and ability to open and close the hand actively
* "Spastic hand and arm" as a prevalent finding verified by clinical examination
* Ability to walk

Exclusion Criteria:

* Musculoskeletal illnesses that affect limbs (e.g., arthrosis, rheumatoid arthritis and amputations).
* BoNT-A treatment of upper limbs in the previous 6 months.
* Orthopedic or neurosurgery procedures performed on the upper limbs in the last 12 months.
* Wrist contracture that prevents patient to play video games
* Severe cognitive deficits
* Other neurological disorders and severe psychiatric illnesses
* Active user of MCVG console at home

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-02-17 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scale score at baseline | Baseline
  Goal Attainment Scale (GAS), where the participant defines specific problem, e.g., activity limitations and participation restrictions caused by upper limb function difficulties, and evaluates to what extent the goal is achieved after treatment and/or training. GAS have previously been utilized to quantify the treatment effects of BoNT-A. Each participant in collaboration with clinicians formulates specific short-term and long-term goals that correspond to the International Classification of Functioning, Disability and Health (ICF) Activity and Participation levels. Minimum scale value -2 (least favorable outcome), Maximum scale value +2 (most favorable outcome)
Goal Attainment Scale score after video games therapy | 3 months after baseline
  Goal Attainment Scale (GAS), where the participant defines specific problem, e.g., activity limitations and participation restrictions caused by upper limb function difficulties, and evaluates to what extent the goal is achieved after treatment and/or training. GAS have previously been utilized to quantify the treatment effects of BoNT-A. Each participant in collaboration with clinicians formulates specific short-term and long-term goals that correspond to the International Classification of Functioning, Disability and Health (ICF) Activity and Participation levels. Minimum scale value -2 (least favorable outcome), Maximum scale value +2 (most favorable outcome)
Goal Attainment Scale score 6 weeks after injection therapy with BoNT-A | 4.5 months after baseline
  Goal Attainment Scale (GAS), where the participant defines specific problem, e.g., activity limitations and participation restrictions caused by upper limb function difficulties, and evaluates to what extent the goal is achieved after treatment and/or training. GAS have previously been utilized to quantify the treatment effects of BoNT-A. Each participant in collaboration with clinicians formulates specific short-term and long-term goals that correspond to the International Classification of Functioning, Disability and Health (ICF) Activity and Participation levels. Minimum scale value -2 (least favorable outcome), Maximum scale value +2 (most favorable outcome)
Goal Attainment Scale score 3 months after injection therapy with BoNT-A | 6 months after baseline
  Goal Attainment Scale (GAS), where the participant defines specific problem, e.g., activity limitations and participation restrictions caused by upper limb function difficulties, and evaluates to what extent the goal is achieved after treatment and/or training. GAS have previously been utilized to quantify the treatment effects of BoNT-A. Each participant in collaboration with clinicians formulates specific short-term and long-term goals that correspond to the International Classification of Functioning, Disability and Health (ICF) Activity and Participation levels. Minimum scale value -2 (least favorable outcome), Maximum scale value +2 (most favorable outcome)
Goal Attainment Scale score at the end of follow up period | 9 months after baseline
  Goal Attainment Scale (GAS), where the participant defines specific problem, e.g., activity limitations and participation restrictions caused by upper limb function difficulties, and evaluates to what extent the goal is achieved after treatment and/or training. GAS have previously been utilized to quantify the treatment effects of BoNT-A. Each participant in collaboration with clinicians formulates specific short-term and long-term goals that correspond to the International Classification of Functioning, Disability and Health (ICF) Activity and Participation levels. Minimum scale value -2 (least favorable outcome), Maximum scale value +2 (most favorable outcome)

SECONDARY OUTCOMES:
Change from baseline Patient Specific Functional Scale score at project defined points of assesment | Baseline, 3 months after baseline, 4,5 months after baseline, 6 months after baseline, 9 months after baseline
  Patient Specific Functional Scale helps participants to define and assess individual goals, motivation and pain related to activities. Scale range 0-10, higher score means a better outcome.
Gross Motor Function Classification System | Baseline
  The Gross Motor Function Classification System or GMFCS is a 5 level clinical classification system that describes the gross motor function of people with cerebral palsy on the basis of self-initiated movement abilities. Classification levels 1-5, lower score means a better outcome
Manual Ability Classification System (MACS) | Baseline
  The Manual Ability Classification System (MACS) describes how patients with cerebral palsy use their hands to handle objects in daily activities. MACS describes five levels. The levels are based on the patient's self-initiated ability to handle objects and their need for assistance or adaptation to perform manual activities in everyday life. Classification levels 1-5, lower score means a better outcome.
Change from baseline Hand Grip Dynamometer score at project defined points of assesment | Baseline, 3 months after baseline, 4,5 months after baseline, 6 months after baseline, 9 months after baseline
  Simultaneous bilateral dynamic grip strength testing With Hand Grip Dynamometer. Score in percentage. The higher the better.
Zancolli Classification Hand Function | Baseline
  This scale explains the grasping and release patterns between the wrist and fingers and hand appearance of the spastic patients. It explains the hand appearance in degrees and that, degrees of extension can be measured using goniometer. The responses of the scale is scored as 1, 1a, 2a, 2b and 3. The best score is 1
House Functional Classification System | Baseline
  Classifies thumb position from 0 to 5. The higher the better.
Change from baseline Modified Ashworth Scales score at project defined points of assesment | Baseline, 3 months after baseline, 4,5 months after baseline, 6 months after baseline, 9 months after baseline
  The Modified Ashworth scale (MAS) measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity. Scale range from 0 to 4, 0 is most favourable outcome.
Change from baseline Range of Motion score at project defined points of assesment | Baseline, 3 months after baseline, 4,5 months after baseline, 6 months after baseline, 9 months after baseline
  Measuring active and passive range of arm joints motion using goniometer
Change from baseline Numeric rating scale (0-10) of symptoms related to pain at 9 months | Baseline, 9 months after baseline
  Self-perceived pain related to spasticity. Score 0 means no pain.
WAIS-IV Coding (Wechsler Adult Intelligence Scale ) | Baseline
  Coding measures visual processing speed, short-term visual memory, and the ability to shift the eyes efficiently back and forth between the "key" and the responses. This task requires fine motor skills but does not require expressive Language. The higher score is better.
Change from baseline Hopkins Symptoms Checklist 25 score at 9 months | Baseline, 9 months after baseline
  The HSCL-25 is a symptom inventory which measures symptoms of anxiety and depression. It consists of 25 items: Part I of the HSCL-25 has 10 items for anxiety symptoms; Part II has 15 items for depression symptoms.
Change from baseline Action Research Arm Test (ARAT) score at project defined points of assesment | Baseline, 3 months after baseline, 4.5 months after baseline, 6 months after baseline, 9 months after baseline
  Assessment for a person's ability to handle objects differing in size, weight and shape. Score range is from 0 to 3, 3 being the best score.
Change from baseline Mini-Balance Evaluation Systems Test score at project defined points of assesment | Baseline, 3 months after baseline, 4.5 months after baseline, 6 months after baseline, 9 months after baseline
  Mini-BESTest includes four subscales: transitions/anticipatory postural control, reactive postural control, sensory orientation and stability in gait. Score range 0 to 28. The higher score the better.
Change from baseline Fatigue Severity Scale (FSS) at 9 months | Baseline, 9 months after baseline
  The Fatigue Severity Scale (FSS) is designed to differentiate fatigue from clinical depression, since both share some of the same symptoms. FSS consists of answering a short questionaire that requires the subject to rate his or her own level of fatigue.
Change from baseline EQ-5D-5L (EuroQol 5 Dimensions 5 Level) Health related quality of life score at 9 months | Baseline, 9 months after baseline
  Descriptive system of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses.

CONTACTS AND LOCATIONS:
Overall Officials: Per Ola Rike, Phd, Study Director — Sunnaas Rehabilitation Hospital

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.